CLINICAL TRIAL: NCT07359118
Title: Evaluation of Healthcare Professionals' Knowledge and Attitudes Regarding Patient-Controlled Analgesia Before and After a Structured Educational Intervention
Brief Title: Assessment of Healthcare Professionals' Knowledge and Attitudes Toward Patient-Controlled Analgesia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2025/04-07
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain Management
Keywords: Patient-Controlled Analgesia; Postoperative Pain; Healthcare Professionals; Education; Knowledge and Attitudes
MeSH Terms: conditions — Pain, Postoperative; Behavior

STUDY DESIGN:
Intervention Model Description: This study uses a non-randomized, parallel-group design. Healthcare professionals assessed before the educational intervention and those assessed after the intervention may not be the same individuals. The pre-education and post-education groups are therefore treated as independent groups, and comparisons are made between these two parallel groups to evaluate the effect of the educational intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Education Assessment Group (Other): Healthcare professionals who complete the study questionnaire before receiving the standardized patient-controlled analgesia educational program.
  Interventions: Behavioral: Patient-Controlled Analgesia Educational Program
- Post-Education Assessment Group (Other): Healthcare professionals who complete the study questionnaire approximately one week after receiving the standardized patient-controlled analgesia educational program.
  Interventions: Behavioral: Patient-Controlled Analgesia Educational Program

INTERVENTIONS:
Behavioral: Patient-Controlled Analgesia Educational Program — A standardized educational program on patient-controlled analgesia delivered to healthcare professionals. The program includes theoretical and practical content covering PCA principles, safe device use, opioid pharmacology, potential complications, patient monitoring, and follow-up. The education is provided through structured sessions and aims to improve participants' knowledge and attitudes regarding PCA.

SUMMARY:
Patient-controlled analgesia (PCA) is a widely used method for postoperative pain management that allows patients to self-administer analgesics according to their pain needs. The safe and effective use of PCA depends largely on the knowledge and awareness of healthcare professionals. Insufficient knowledge may lead to improper use of PCA devices and increase the risk of complications affecting patient safety.

The aim of this study will be to evaluate healthcare professionals' knowledge and attitudes regarding patient-controlled analgesia and to assess the effect of a structured educational intervention on these outcomes. This interventional, pre-post comparative study will be conducted among healthcare professionals working in surgical clinics, operating rooms, and intensive care units at a tertiary care hospital.

Participants will complete a structured questionnaire assessing demographic characteristics, PCA-related knowledge, and attitudes before receiving a standardized educational program on patient-controlled analgesia. The same questionnaire will be administered again one week after the education. Changes in knowledge and attitude scores before and after the educational intervention will be analyzed using appropriate statistical methods.

DETAILED DESCRIPTION:
Patient-controlled analgesia (PCA) is an important component of postoperative pain management that allows patients to self-administer analgesic medications within predetermined safety limits. The effectiveness and safety of PCA depend not only on appropriate device programming and pharmacological selection but also on the knowledge, awareness, and clinical practices of healthcare professionals responsible for patient education, monitoring, and device management.

This study will be designed as a semi-experimental, interventional, pre-post comparative study to evaluate healthcare professionals' knowledge and attitudes regarding patient-controlled analgesia and to assess the impact of a structured educational intervention on these outcomes. The study will be conducted among healthcare professionals working in surgical wards, operating rooms, and intensive care units of a tertiary care hospital.

Eligible participants will include physicians, nurses, anesthesia technicians, and midwives aged 18 years and older who are actively involved in perioperative patient care. Healthcare professionals who decline participation, do not complete the questionnaires, or are not working in the specified clinical units will be excluded from the study.

Before the educational intervention, participants will complete a structured questionnaire consisting of three sections. The first section will collect demographic and professional information, including age, sex, profession, years of clinical experience, department of employment, and previous experience with PCA-treated patients. The second section will assess knowledge related to patient-controlled analgesia using 32 true/false items covering PCA principles, routes of administration, device characteristics, opioid analgesics, contraindications, complications, device management, and patient monitoring. The third section will evaluate attitudes toward PCA using 28 statements rated on a four-point Likert scale ranging from "strongly disagree" to "strongly agree."

Following baseline assessment, a standardized educational program on patient-controlled analgesia will be delivered to all participants. The educational content will include theoretical and practical information on PCA principles, safe device use, opioid pharmacology, complication recognition, and patient follow-up. One week after completion of the educational intervention, the same questionnaire will be re-administered under identical conditions.

Changes in knowledge and attitude scores before and after the educational intervention will be analyzed using appropriate statistical methods to determine the effect of education on healthcare professionals' understanding and perceptions of patient-controlled analgesia. The findings of this study are expected to contribute to improved patient safety and quality of postoperative pain management by highlighting the importance of structured educational programs for healthcare professionals involved in PCA practices.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare professionals (physicians, nurses, anesthesia technicians, and midwives) working in surgical wards, operating rooms, or intensive care units.
* Aged 18 years or older.
* Actively involved in perioperative patient care.
* Willing to participate in the study and provide informed consent.

Exclusion Criteria:

* Healthcare professionals who decline to participate.
* Incomplete or missing questionnaire responses.
* Healthcare professionals not working in the specified clinical units.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Change in Knowledge Score on Patient-Controlled Analgesia | From baseline (pre-education) to 1 week after the educational intervention
  The primary outcome is the change in healthcare professionals' knowledge regarding patient-controlled analgesia, assessed using a structured questionnaire consisting of true/false items administered before and after the educational intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Kütahya City Hospital, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Song Z, Cai J, Zhou Y, Jiang Y, Huang S, Gu L, Tan J. Knowledge, Attitudes and Practices Among Anesthesia and Thoracic Surgery Medical Staff Toward Ai-PCA. J Multidiscip Healthc. 2024 Jul 10;17:3295-3304. doi: 10.2147/JMDH.S468539. eCollection 2024. PMID 39006875
- [Background] Kang MR, Kwon YJ. Nurses' knowledge and attitudes toward patient-controlled analgesia for postoperative pain control in a tertiary hospital in South Korea. BMC Nurs. 2022 Nov 22;21(1):319. doi: 10.1186/s12912-022-01106-7. PMID 36419116
- [Background] Chen YR, Chen CC, Wu WW, Tang FI, Lu LC. Nurses' knowledge of and attitude toward postoperative patient-controlled analgesia (PCA) and the associated factors. BMC Nurs. 2024 Jan 5;23(1):21. doi: 10.1186/s12912-024-01702-9. PMID 38183011